CLINICAL TRIAL: NCT05207163
Title: Continuing Medical Education (CME) Intervention to Improve Knowledge About Viral Hepatitis B-C: A Randomized Controlled Trial Pilot at Primary-level Hospitals in Ho Chi Minh City
Brief Title: Continuing Medical Education to Improve Knowledge of Viral Hepatitis B-C in Primary Healthcare Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Pham Ngoc Thach University of Medicine (Other)
Responsible Party: Principal Investigator, Le Hong Duc, Lecturer - Researcher, Pham Ngoc Thach University of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 511/TĐHYKPNT-HĐĐĐ
Record Dates: First submitted 2021-12-09; First posted 2022-01-26 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Viral Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Received CME (Experimental)
  Interventions: Behavioral: Continuing medical education
- Not received CME (No Intervention)

INTERVENTIONS:
Behavioral: Continuing medical education — Education section about knowledge of transmissions, severity of viral hepatitis B-C and update treatment strategy of the HBV-HCV
  Arms: Received CME

SUMMARY:
The purpose of study is identifying the effectiveness of 'continuing medical education' (CME) to primary healthcare worker to improve knowledge about viral hepatitis B-C

ELIGIBILITY:
Inclusion Criteria:

* Currently working at Outpatient department, Primary-level hospitals
* Having Practicing Certificate
* Not attending any long-term education
* Accepting ICF

Exclusion Criteria:

* Not attending the full number of lessons
* Not answering the questionnaire

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-02-10 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in Test Scores on Knowledge about Hepatitis B-C from Baseline to 6 months | 6 months
  Participants have exams pre- and post-6-months-course, which is multiple choice questions. The test score is average number of correct answers. The pre- and post-6-months exams use the same structure and questions. A change in test score is the difference between test score of the post-6-months-exam and test score of the pre-course-exam.

CONTACTS AND LOCATIONS:
Overall Officials: Lê H Đức, Medicine, Principal Investigator — Pham Ngoc Thach University of Medicine
Locations (1):
- Lê Hồng Đức, Tháng 07, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided